CLINICAL TRIAL: NCT03790085
Title: Identification of Multi-modal Bio-markers for Early Diagnosis and Treatment Prediction in Schizophrenia Individuals
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Shanghai Mental Health Center (Other); Nanjing Medical University (Other); Tianjin Anding Hospital (Other); Harbin First Specialist Hospital (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); Anhui Mental Health Center (Unknown); Wuhan Psychiatric Hospital (Unknown); Wenzhou Seventh People's Hospital (Other Government); First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Chunshui Yu, Vice president of Tianjin Medical University, Tianjin Medical University General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018YFC1314300
Record Dates: First submitted 2018-12-25; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Schizophrenia; Major Depressive Disorder; Anxiety Disorders
Keywords: Precision medicine; Bio-marker; Neuroimaging; Molecular genetics; Neurobiochemical; Early diagnosis; Early prediction
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Anxiety Disorders; Disease | interventions — Risperidone; Olanzapine; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Risperidone (Experimental): It can be used after schizophrenia is diagnosed. Risperidone affects prolactin and may affect menstruation in young women, so we will try not to use it in such patients. Patients were randomized to a single Risperidone control trial for 8 weeks to evaluate the clinical efficacy of the patients. Risperidone routine daily 2-6 mg, up to 8 mg, can be taken orally twice a day.
  Interventions: Drug: Risperidone
- Olanzapine (Experimental): It can be used after schizophrenia is diagnosed. Olanzapine is not generally used in patients with diabetes and hyperlipidemia. Patients were randomized to a single Olanzapine control trial for 8 weeks to evaluate the clinical efficacy of the patients. Olanzapine is available once or twice a day, starting at 5 mg daily and up to 20 mg daily.
  Interventions: Drug: Olanzapine
- Aripiprazole (Experimental): It can be used after schizophrenia is diagnosed. Aripiprazole has no specific contraindications. Patients were randomized to a single Aripiprazole control trial for 8 weeks to evaluate the clinical efficacy of the patients. Aripiprazole is taken orally once a day, starting at 10 mg daily and up to 30 mg daily.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Risperidone — Risperidone tablet
  Arms: Risperidone
Drug: Olanzapine — Olanzapine tablet
  Arms: Olanzapine
Drug: Aripiprazole — Aripiprazole tablet
  Arms: Aripiprazole

SUMMARY:
This study aims to screen and validate multi-scale bio-markers for early diagnosis and medication monitoring for early schizophrenia, including the genetic, neurobiochemistry, neuroimaging and eletrophysiological measures. Based on the validated bio-markers, the present study further tries to build several prediction models for early differential diagnosis of schizophrenia from healthy controls and other mental diseases (such as the major depression and anxiety disorders), biological sub-typing and diagnosis of the schizophrenia sub-types, and early prediction of the medication effects.

DETAILED DESCRIPTION:
Schizophrenia is one of the most important diseases that threaten the health of Chinese people. In view of the current lack of objective biological markers in the diagnosis and treatment of schizophrenia, as well as the lack of effective early diagnosis methods and curative effect prediction methods, the investigators carried out joint research by integrating research teams from molecular genetics, neurobiochemistry, psychiatry, medical imaging, information science and other fields. The overall objective of the project is to establish a bio-marker system for individualized diagnosis and treatment of early schizophrenia. Specific research contents include: screening and verifying multidimensional objective biological markers such as genetics, neurobiochemistry, neuroimaging, electrophysiology, which is related to early diagnosis and efficacy prediction of schizophrenia through big data analysis of healthy controls and patients with first episode schizophrenia, depression and anxiety disorder. Pattern recognition method is used to build the individualized early diagnosis model, biological sub-type clustering model, biological sub-type individualized diagnosis model and early curative effect prediction model of schizophrenia. Based on the individualized diagnosis and treatment prediction model of schizophrenia, the individualized diagnosis and treatment toolkit was developed, and the individualized diagnosis and treatment prediction cloud platform was established to provide assist for clinicians.

ELIGIBILITY:
Inclusion Criteria for patients:

* According with American mental disorder diagnosis and Diagnostic criteria for schizophrenia, major depressive disorder, and anxiety disorder in the statistical manual DSM-IV
* The time from the onset of symptoms for the first time to participate in study is less than 12 months
* No any anti-psychotic drugs or medication was taken more than 14 days
* Han nationality
* 18 to 45 years old
* Right-handed

Inclusion Criteria for healthy controls:

* Han nationality
* Right-handedness
* Gender, age and education level are matched with patients
* 18 to 45 years old
* Any mental disorder diagnosis in DSM-IV was excluded
* There were no relatives with severe mental disorder in the two or three generations

Exclusion Criteria:

* The patient has other psychiatric disorder beside the illness
* A history of psychoactive substance use, accompanied by severe physical disease
* Have a history of epilepsy or coma
* Women who are pregnant or breast-feeding
* Accompanied by metal implants, claustrophobia and other contraindications of MRI scan

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2700 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 30-45 minutes
  It is a scale involved and standardized for assessing the severity of symptoms of different types of schizophrenia. Of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale. Each of the 30 items is accompanied by a specific definition as well as detailed anchoring criteria for all seven rating points. The scores for these scales are arrived at by summation of ratings across component items. These seven points represent increasing levels of psychopathology, as follows: 1- absent, 2- minimal, 3-mild, 4-moderate, 5-moderate severe, 6-severe, 7-extreme. Therefore, the potential ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale. A rating of 7 (extreme) refers to the most serious level of psychopathology in each item, so the higher the score is, the more serious the physical level is.
Clinical Global Impression(CGI) | 10-15 minutes
  the CGI is a 3-item observer-rated scale that measures illness severity (CGIS), global improvement or change (CGIC) and therapeutic response.The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Treatment response ratings should take account of both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side-effects) and 4 (unchanged or worse and side-effects outweigh the therapeutic effects). Each component of the CGI is rated separately; the instrument does not yield a global score.

CONTACTS AND LOCATIONS:
Overall Officials: Chunshui Yu, MD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gusev A, Mancuso N, Won H, Kousi M, Finucane HK, Reshef Y, Song L, Safi A; Schizophrenia Working Group of the Psychiatric Genomics Consortium; McCarroll S, Neale BM, Ophoff RA, O'Donovan MC, Crawford GE, Geschwind DH, Katsanis N, Sullivan PF, Pasaniuc B, Price AL. Transcriptome-wide association study of schizophrenia and chromatin activity yields mechanistic disease insights. Nat Genet. 2018 Apr;50(4):538-548. doi: 10.1038/s41588-018-0092-1. Epub 2018 Apr 9. PMID 29632383
- [Result] Zhu J, Zhuo C, Xu L, Liu F, Qin W, Yu C. Altered Coupling Between Resting-State Cerebral Blood Flow and Functional Connectivity in Schizophrenia. Schizophr Bull. 2017 Oct 21;43(6):1363-1374. doi: 10.1093/schbul/sbx051. PMID 28521048
- [Result] Drysdale AT, Grosenick L, Downar J, Dunlop K, Mansouri F, Meng Y, Fetcho RN, Zebley B, Oathes DJ, Etkin A, Schatzberg AF, Sudheimer K, Keller J, Mayberg HS, Gunning FM, Alexopoulos GS, Fox MD, Pascual-Leone A, Voss HU, Casey BJ, Dubin MJ, Liston C. Resting-state connectivity biomarkers define neurophysiological subtypes of depression. Nat Med. 2017 Jan;23(1):28-38. doi: 10.1038/nm.4246. Epub 2016 Dec 5. PMID 27918562
- [Result] Jaffe AE, Gao Y, Deep-Soboslay A, Tao R, Hyde TM, Weinberger DR, Kleinman JE. Mapping DNA methylation across development, genotype and schizophrenia in the human frontal cortex. Nat Neurosci. 2016 Jan;19(1):40-7. doi: 10.1038/nn.4181. Epub 2015 Nov 30. PMID 26619358
- [Result] Marshall CR, Howrigan DP, Merico D, Thiruvahindrapuram B, Wu W, Greer DS, Antaki D, Shetty A, Holmans PA, Pinto D, Gujral M, Brandler WM, Malhotra D, Wang Z, Fajarado KVF, Maile MS, Ripke S, Agartz I, Albus M, Alexander M, Amin F, Atkins J, Bacanu SA, Belliveau RA Jr, Bergen SE, Bertalan M, Bevilacqua E, Bigdeli TB, Black DW, Bruggeman R, Buccola NG, Buckner RL, Bulik-Sullivan B, Byerley W, Cahn W, Cai G, Cairns MJ, Campion D, Cantor RM, Carr VJ, Carrera N, Catts SV, Chambert KD, Cheng W, Cloninger CR, Cohen D, Cormican P, Craddock N, Crespo-Facorro B, Crowley JJ, Curtis D, Davidson M, Davis KL, Degenhardt F, Del Favero J, DeLisi LE, Dikeos D, Dinan T, Djurovic S, Donohoe G, Drapeau E, Duan J, Dudbridge F, Eichhammer P, Eriksson J, Escott-Price V, Essioux L, Fanous AH, Farh KH, Farrell MS, Frank J, Franke L, Freedman R, Freimer NB, Friedman JI, Forstner AJ, Fromer M, Genovese G, Georgieva L, Gershon ES, Giegling I, Giusti-Rodriguez P, Godard S, Goldstein JI, Gratten J, de Haan L, Hamshere ML, Hansen M, Hansen T, Haroutunian V, Hartmann AM, Henskens FA, Herms S, Hirschhorn JN, Hoffmann P, Hofman A, Huang H, Ikeda M, Joa I, Kahler AK, Kahn RS, Kalaydjieva L, Karjalainen J, Kavanagh D, Keller MC, Kelly BJ, Kennedy JL, Kim Y, Knowles JA, Konte B, Laurent C, Lee P, Lee SH, Legge SE, Lerer B, Levy DL, Liang KY, Lieberman J, Lonnqvist J, Loughland CM, Magnusson PKE, Maher BS, Maier W, Mallet J, Mattheisen M, Mattingsdal M, McCarley RW, McDonald C, McIntosh AM, Meier S, Meijer CJ, Melle I, Mesholam-Gately RI, Metspalu A, Michie PT, Milani L, Milanova V, Mokrab Y, Morris DW, Muller-Myhsok B, Murphy KC, Murray RM, Myin-Germeys I, Nenadic I, Nertney DA, Nestadt G, Nicodemus KK, Nisenbaum L, Nordin A, O'Callaghan E, O'Dushlaine C, Oh SY, Olincy A, Olsen L, O'Neill FA, Van Os J, Pantelis C, Papadimitriou GN, Parkhomenko E, Pato MT, Paunio T; Psychosis Endophenotypes International Consortium; Perkins DO, Pers TH, Pietilainen O, Pimm J, Pocklington AJ, Powell J, Price A, Pulver AE, Purcell SM, Quested D, Rasmussen HB, Reichenberg A, Reimers MA, Richards AL, Roffman JL, Roussos P, Ruderfer DM, Salomaa V, Sanders AR, Savitz A, Schall U, Schulze TG, Schwab SG, Scolnick EM, Scott RJ, Seidman LJ, Shi J, Silverman JM, Smoller JW, Soderman E, Spencer CCA, Stahl EA, Strengman E, Strohmaier J, Stroup TS, Suvisaari J, Svrakic DM, Szatkiewicz JP, Thirumalai S, Tooney PA, Veijola J, Visscher PM, Waddington J, Walsh D, Webb BT, Weiser M, Wildenauer DB, Williams NM, Williams S, Witt SH, Wolen AR, Wormley BK, Wray NR, Wu JQ, Zai CC, Adolfsson R, Andreassen OA, Blackwood DHR, Bramon E, Buxbaum JD, Cichon S, Collier DA, Corvin A, Daly MJ, Darvasi A, Domenici E, Esko T, Gejman PV, Gill M, Gurling H, Hultman CM, Iwata N, Jablensky AV, Jonsson EG, Kendler KS, Kirov G, Knight J, Levinson DF, Li QS, McCarroll SA, McQuillin A, Moran JL, Mowry BJ, Nothen MM, Ophoff RA, Owen MJ, Palotie A, Pato CN, Petryshen TL, Posthuma D, Rietschel M, Riley BP, Rujescu D, Sklar P, St Clair D, Walters JTR, Werge T, Sullivan PF, O'Donovan MC, Scherer SW, Neale BM, Sebat J; CNV and Schizophrenia Working Groups of the Psychiatric Genomics Consortium. Contribution of copy number variants to schizophrenia from a genome-wide study of 41,321 subjects. Nat Genet. 2017 Jan;49(1):27-35. doi: 10.1038/ng.3725. Epub 2016 Nov 21. PMID 27869829
- [Derived] Lei X, Ren J, Teng X, Guo C, Wu Z, Yu L, Chen X, Fu L, Zhang R, Wang D, Chen Y, Zhang Y, Zhang C. Characterizing Unipolar and Bipolar Depression by Alterations in Inflammatory Mediators and the Prefrontal-Limbic Structural Network. Depress Anxiety. 2023 May 24;2023:5522658. doi: 10.1155/2023/5522658. eCollection 2023. PMID 40224600
- [Derived] Fu L, Ren J, Lei X, Wang Y, Chen X, Zhang R, Li Q, Teng X, Guo C, Wu Z, Yu L, Wang D, Chen Y, Qin J, Yuan A, Zhang C. Association of anhedonia with brain-derived neurotrophic factor and interleukin-10 in major depressive disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2024 Jul 13;133:111023. doi: 10.1016/j.pnpbp.2024.111023. Epub 2024 May 1. PMID 38701878
- [Derived] Lei X, Fang X, Ren J, Teng X, Guo C, Wu Z, Yu L, Wang D, Chen Y, Zhou Y, Wu Y, Zhang Y, Zhang C. Plasma Apo-E mediated corticospinal tract abnormalities and suicidality in patients with major depressive disorder. Eur Arch Psychiatry Clin Neurosci. 2024 Aug;274(5):1167-1175. doi: 10.1007/s00406-023-01749-w. Epub 2024 Jan 24. PMID 38265467